CLINICAL TRIAL: NCT05160805
Title: A Phase 1b Multicenter, Randomized, Single-Masked, Sham-Controlled Study of the Safety and Tolerability of ONL1204 Ophthalmic Solution in Patients with Progressing Open Angle Glaucoma
Brief Title: A Phase 1b Study of ONL1204 Ophthalmic Solution in Patients with Progressing Open Angle Glaucoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ONL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONL1204-OAG-001
Record Dates: First submitted 2021-12-06; First posted 2021-12-16 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Open Angle Glaucoma
Keywords: Progressing; Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment Group A (Experimental): ONL1204 Ophthalmic solution (Dose A) administered by intravitreal injection
  Interventions: Drug: ONL1204 Ophthalmic solution (Dose A)
- Treatment Group B (Experimental): ONL1204 Ophthalmic solution (Dose B) administered by intravitreal injection
  Interventions: Drug: ONL1204 Ophthalmic solution (Dose B)
- Treatment Group C (Sham Comparator): Sham procedure without penetrating the eye
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Drug: ONL1204 Ophthalmic solution (Dose A) — Liquid formulation administered by intravitreal (IVT) injection
  Arms: Treatment Group A
Drug: ONL1204 Ophthalmic solution (Dose B) — Liquid formulation administered by intravitreal (IVT) injection
  Arms: Treatment Group B
Procedure: Sham procedure — A sham procedure looks like a real injection into the eye but does not penetrate the eye and it does not have any study drug. The procedure is done by touching the eye surface with a syringe without a needle.
  Arms: Treatment Group C

SUMMARY:
The purpose of this study is to demonstrate the safety and tolerability of ONL1204 Ophthalmic Solution in patients with progressing open angle glaucoma.

ONL1204 Ophthalmic Solution is a first-in-class inhibitor of fragment apoptosis stimulator (Fas) receptor-mediated cell death that has demonstrated protection of multiple retinal cell types in numerous preclinical models of retinal disease. Apoptosis of retinal ganglion cells is associated with progressive glaucoma. Nonclinical data on ONL1204 Ophthalmic Solution suggest that ONL1204 Ophthalmic Solution may inhibit the cell death pathways in these cells.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥18 years old
2. Able and willing to give informed consent and attend study visits
3. Controlled intraocular pressure (IOP) (≤21 mmHg) in both eyes for all previous 3 visits before Screening and at Screening in both eyes
4. Prior to screening, 3 or more Humphrey Visual Field (HVF) tests (with acceptable reliability standards) or 3 or more Optical Coherence Tomography (OCT) studies of the study eye on record
5. Open angle glaucoma that is progressing in the study eye
6. HVF 24-2 at Screening with acceptable reliability standards and MD scores

Exclusion Criteria:

Considerations for either eye

1. Best Corrected Visual Acuity (BCVA) at Screening of ≤64 letters (Snellen equivalent of worse than 20/50)
2. Severe open angle glaucoma
3. Glaucoma due to non-open angle causes
4. Worse than mild non-proliferative diabetic retinopathy

   Considerations for study eye:
5. Visual field results suggestive of another disease (eg, altitudinal field defect)
6. Evidence of macular edema based on OCT imaging and Investigator's judgement
7. Previous intravitreal (IVT) injections, history of retinal surgery, history of retinal laser
8. Cataract surgery within 3 months of Screening or yttrium-aluminum-garnet capsulotomy (YAG) within 4 weeks of Screening
9. Anticipated need for surgical or procedural intervention for glaucoma, cataract, posterior capsular opacity, refractive error, or retinal conditions during the study

   Other general exclusion criteria:
10. The requirement for oral carbonic anhydrase inhibitors to control intraocular pressure
11. Severe, unstable, or uncontrolled cardiovascular, diabetic, renal, or pulmonary disease, based on Investigator's judgement
12. Systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg
13. Women who are pregnant, breastfeeding, or contemplating pregnancy during the study period and men who are contemplating contributing sperm for a biologic child during the study period
14. Participation in other ophthalmic clinical trials or use of any other investigational drugs or devices in either eye or systemically for 3 months before Screening (Visit 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of ONL1204 as assessed by AE reporting and clinical evaluations | up to 39 weeks
  Adverse event reporting, ophthalmic examination to evaluate the anterior and posterior segments of the eye, best-corrected visual acuity, intraocular pressure, electroretinogram, vital signs, clinical laboratory evaluations, and ophthalmic imaging results

CONTACTS AND LOCATIONS:
Locations (11):
- Australia (9):
  - Albury Eye Clinic Wodonga, Albury, New South Wales
  - Sydney Eye Surgeons, Hurstville, New South Wales
  - PersonalEYES, Parramatta, New South Wales
  - Eye Associates, Sydney, New South Wales
  - Armadale Eye Clinic, Armadale, Victoria
  - Melbourne Eye Specialists, Fitzroy, Victoria
  - North West Eye Specialists, Gladstone Park, Victoria
  - Centre for Eye Research Australia (CERA), Melbourne, Victoria
  - Waverely Eye Clinic, Waverley, Victoria
- New Zealand (2):
  - Eye Institute Limited, Remuera, Auckland
  - Capital Eye Specialists, Wellington, Wellington Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ONL Therapeutics corporate website — https://www.onltherapeutics.com/clinical-trials/